CLINICAL TRIAL: NCT01185795
Title: Efficacy of a Microencapsulated Probiotic Yogurt Formulation as a Health Promoting Agent
Brief Title: Efficacy of Cardioviva™ Probiotic Yogurt Formulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Micropharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-001
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Hypercholesterolemia
Keywords: yogurt; probiotic; cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardioviva™ yogurt (Experimental)
  Interventions: Dietary Supplement: Cardioviva™ yogurt
- Placebo yogurt (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo yogurt

INTERVENTIONS:
Dietary Supplement: Cardioviva™ yogurt — L. reuteri cardioviva in yogurt, twice per day (BID), 6 weeks
  Arms: Cardioviva™ yogurt
Dietary Supplement: Placebo yogurt — yogurt, twice per day (BID), 6 weeks
  Arms: Placebo yogurt

SUMMARY:
Background: Several studies have reported limited or no reduction in serum lipid concentrations in response to probiotic formulations. More recently, probiotics have shown promise in treating metabolic disease, due to improved strain selection and delivery technologies.

Objective: To evaluate the lipid lowering efficacy of a yogurt formulation containing microencapsulated Bile Salt Hydrolase (BSH)-active Lactobacillus reuteri cardioviva, taken twice per day over 6 weeks, in subjects with hypercholesterolemia.

Design: This is a double-blinded, multi-centric, placebo-controlled, randomized, parallel-arm study. The study will last a total of 10 weeks including 2-week wash-out, 2-week run-in, and 6- week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females.
* Aged 18-74 years old.
* Low Density Lipoprotein (LDL-C) above 3.4 mmol/L (<15% variation between visits V1 and V2-1).
* Triglyceride (TG) levels below 4.0 mmol/l (check at V0 and V2-1).
* Body Mass Index (BMI) range was 22 to 32 kg/m2.
* Ability to understand dietary procedures.
* Judged by the investigators as compliant (>80%) with product consumption (check at V2-1), and motivated.
* Signed informed consent form prior to inclusion in the study
* Note: Subjects were permitted to take stable doses of thyroid hormone, anti-hypertensive agents, and contraceptive hormones (e.g. contraceptive pills or patches), as long as these were continued equivalently throughout the duration of study.

Exclusion Criteria:

* Use of statin or other cholesterol lowering prescription drugs within the last 6 months.
* Use of plant sterols, omega-3, fish oil, soy protein, soluble oat fiber, psyllium seed husk, or other cholesterol lowering non-prescription supplements within last 3 months.
* History of chronic use of alcohol (>2 drinks/day).
* Use of systemic antibodies, corticosteroids, androgens, or phenytoin.
* Myocardial infarction, coronary artery bypass, or other major surgical procedures within the last six months.
* Lactose intolerance or allergies to dairy products.
* History of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, diabetes, gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer (evidence of active lesions, chemotherapy or surgery in the past year).
* Chronic user of probiotics or fiber laxative (greater than 2 doses/week), or stimulant laxatives.
* History of eating disorders.
* Exercise greater than 15 miles/week or 4,000 kcal/week.
* Pregnancy, breast feeding, or intent to get pregnant.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be the percent change from baseline in Low Density Lipoprotein Cholesterol (LDL-C) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell L Jones, MD, MEng, Study Director — Micropharma Limited